CLINICAL TRIAL: NCT00696605
Title: Assessment of Circulating Copeptin Levels in Healthy Subjects and Patients With Renal Insufficiency After Oral Water Load and Hypertonic Saline Infusion
Status: Completed | Type: Observational
Sponsor: Hospital Centre Biel/Bienne (Other)
Collaborators: Brahms AG (Industry)
Responsible Party: Principal Investigator, Jonas Rutishauser, M.D., Hospital Centre Biel/Bienne
Other Study IDs: Swiss AVP-Copeptin Trial
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Hypoosmolality; Hyperosmolality; Renal Failure
Keywords: Hypoosmolality; Hyperosmolality; Copeptin; Vasopressin
MeSH Terms: conditions — Renal Insufficiency; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The are 2 principal goals in this study:

1. To measure plasma copeptin levels in healthy subjects and to correlate them with plasma AVP concentrations and urine osmolalities in iso-, hypo-, and hyperosmolar states.
2. To measure plasma copeptin concentrations in patients with chronic renal failure under the same conditions described above, in order to characterize the impact of renal function on circulating copeptin levels in correlation to plasma AVP and urine osmolality.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure grade I through IV
* healthy age-matched controls

Exclusion Criteria:

* chronic renal failure grade V
* heart failure
* liver disease
* nephrotic syndrome
* anemia (hemoglobin level < 100 g/L)
* uncontrolled hypertension (systolic BP > 160 mmHg; diastolic BP > 95 mm Hg)
* coexisting severe disease
* known thyroid disease
* known hypocortisolism
* known hypercortisolism
* known diabetes insipidus
* pregnancy
* lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers; patients with chronic renal failure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Internal Medicine, Hospital Center, Biel/Bienne, Switzerland

REFERENCES:
- [Derived] Balanescu S, Kopp P, Gaskill MB, Morgenthaler NG, Schindler C, Rutishauser J. Correlation of plasma copeptin and vasopressin concentrations in hypo-, iso-, and hyperosmolar States. J Clin Endocrinol Metab. 2011 Apr;96(4):1046-52. doi: 10.1210/jc.2010-2499. Epub 2011 Feb 2. PMID 21289257